CLINICAL TRIAL: NCT03754153
Title: Phase 2a Two-site Randomised Controlled Trial to Determine Safety of and Adherence With a New 'Binocularly Balanced Viewing' Treatment for Unilateral Amblyopia Compared With Standard Treatment in Children Age 3-8 Years
Brief Title: Binocularly Balanced Viewing Study
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DALA1031
Record Dates: First submitted 2017-07-31; First posted 2018-11-27 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: Two-group parallel randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: At each site, a masked orthoptist will carry out the study assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balanced Binocular Viewing (BBV) (Experimental): The experimental intervention will be BBV treatment, i.e. viewing movies for one hour or 2x30min/day on a Nintendo 3DSXL console. With this technology, the Investigators will show blurred images to the better-seeing eye and normal images to the amblyopic eye, encouraging the use of the amblyopic eye and improving acuity.
  Interventions: Device: Balanced Binocular Viewing (BBV)
- Standard Therapy - Occlusion (patching) or blurring (atropine) (Active Comparator): The control intervention will be either atropine eyedrops twice a week or daily occlusion (patching) therapy of the better-seeing eye (which are the current standards). As per clinical standard, parents will be offered the choice of occlusion or eyedrop treatment.
  Interventions: Other: Standard Therapy - Occlusion (patching) or blurring (atropine)

INTERVENTIONS:
Device: Balanced Binocular Viewing (BBV) — The dose of BBV therapy will be one hour a day or 2x30 min/day (depending on child's attention span and/or need to implement the treatment around the family daily routine).
  Arms: Balanced Binocular Viewing (BBV)
Other: Standard Therapy - Occlusion (patching) or blurring (atropine) — The prescribed dose of occlusion treatment / patching (parental choice) will depend on the severity of amblyopia, as by current clinical practice based on PEDIG studies
  Arms: Standard Therapy - Occlusion (patching) or blurring (atropine)

SUMMARY:
Amblyopia is treated by glasses and patches or blurring eyedrops to the good eye. This works in about 70% of children, but parents and children strongly dislike these treatments which may carry on for years and involve frequent clinic visits. In this pilot trial, 66 children will receive, at random, either a Nintendo 3DSXL console with movies, or standard patching/blurring eye-drop treatment. The Investigators will monitor adverse events (double vision), change in the balance between the two eyes and in visual acuity over 16 weeks.

DETAILED DESCRIPTION:
"Lazy eye" (amblyopia) is the commonest sight problem in children, affecting about one in 30 children. It is caused by a difference in spectacle prescription between the eyes and/or a squint (eye misalignment), with the brain ignoring one eye. Amblyopia is treated by glasses and patches or blurring eyedrops to the good eye. This works in about 70% of children, but parents and children strongly dislike these treatments which may carry on for years and involve frequent clinic visits.

The Investigators have developed an exciting new treatment: children watch customized movies for an hour a day on a hand-held 3D computer-game console. The Investigators blur the picture that the good eye sees to match it with what the weaker eye sees. They have tested this approach on 22 children, with an average improvement in vision by three lines on the test chart over 8 - 24 weeks, which may be faster than with standard treatment. Parents and children the Investigators have spoken with like both the idea of research in this area and the engaging nature of this device. The Investigators now need to assess how the new treatment compares with standard treatment, but first need to ensure that the new treatment is safe and that families will use it.

In this pilot trial, 66 children will receive, at random, either a Nintendo 3DSXL console with movies, or standard patching/blurring eye-drop treatment. The Investigators will monitor adverse events (double vision), change in the balance between the two eyes and in visual acuity over 16 weeks. Parents and children have helped develop this pilot - this involvement will be continued throughout the study. At study completion, children and parents will be involved in deciding how best to communicate the findings on hospital websites, in newsletters, at conferences and in medical journals.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3.0 and less than 8.0 years
* unilateral anisometropic, strabismic or combined mechanism amblyopia
* best-corrected crowded logMAR visual acuity (BCVA) in the amblyopic eye worse than 0.2logMar
* best corrected visual acuity in the better seeing eye 0.2 or better
* difference in best corrected visual acuity between the two eyes of 0.2 logMAR or more
* adapted to spectacles with no improvement in acuity in affected eye for two consecutive visits
* no previous treatment for amblyopia other than glasses

Exclusion Criteria:

* ocular cause for reduced visual acuity
* inability to co-operate with assessment tests
* other developmental disorders or learning or neurological disability that would impact on adherence to treatment
* photopic epilepsy
* myopia with spherical equivalent of greater than -6.00DS
* previous intraocular surgery
* inability to perform a crowded letter logMAR visual acuity test using a clinical trials standard testing method (ATS-HOTV protocol), either by naming or by matching letters

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The evaluation of safety of the experimental intervention | 16 weeks from randomization
  To measure changes in suppression/interocular balance (considered to precede double vision) at 16 weeks from baseline, using a novel test of interocular balance, a contrast-sensitivity test presented on a PC

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Dahlmann-Noor, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual-level data will be made available on request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Will be made available after publication of the trial findings.
Access Criteria: As per review by sponsor and principal investigator.

REFERENCES:
- [Derived] Dahlmann-Noor AH, Greenwood JA, Skilton A, Baker D, Abbas M, Clay E, Khandelwal P, Dunham D, Ludden S, Davis A, Dehbi HM, Dakin SC. Feasibility of a new 'balanced binocular viewing' treatment for unilateral amblyopia in children aged 3-8 years (BALANCE): results of a phase 2a randomised controlled feasibility trial. BMJ Open. 2024 Jul 30;14(7):e082472. doi: 10.1136/bmjopen-2023-082472. PMID 39079927
- [Derived] Dahlmann-Noor AH, Greenwood JA, Skilton A, Baker D, Ludden S, Davis A, Dehbi HM, Dakin SC. Phase 2a randomised controlled feasibility trial of a new 'balanced binocular viewing' treatment for unilateral amblyopia in children age 3-8 years: trial protocol. BMJ Open. 2022 May 24;12(5):e051423. doi: 10.1136/bmjopen-2021-051423. PMID 35613759